CLINICAL TRIAL: NCT06243198
Title: A Phase 1, Participant- and Investigator-blinded, Randomized, Single-dose Study to Investigate the Safety and Pharmacokinetics of Lebrikizumab in Healthy Chinese Participants
Brief Title: A Study to Investigate the Safety and Pharmacokinetics of Lebrikizumab in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 18791; J2T-MC-KGBV (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Safety; Lebrikizumab; Chinese
MeSH Terms: interventions — lebrikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 250 mg Lebrikizumab (Experimental): Participants received single dose of 250 milligram (mg) lebrikizumab administered as subcutaneous (SC) injection on day 1.
  Interventions: Drug: Lebrikizumab
- 500 mg Lebrikizumab (Experimental): Participants received single dose of 500 mg lebrikizumab administered as SC injection on day 1.
  Interventions: Drug: Lebrikizumab
- Placebo (Placebo Comparator): Participants received single dose of placebo administered as SC injection on day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lebrikizumab — Administered subcutaneously (SC)
  Other Names: LY3650150
  Arms: 250 mg Lebrikizumab; 500 mg Lebrikizumab
Drug: Placebo — Administered subcutaneously (SC)
  Arms: Placebo

SUMMARY:
The main purpose of this study is to determine the tolerability and side effects related to lebrikizumab comparing with placebo given as a single dose administered under the skin to healthy Chinese participants. The study will also assess how fast lebrikizumab gets into the blood stream and how long the body takes to get rid of it. Each enrolled participant will receive a single dose of either Lebrikizumab or placebo.

For each participant, the total duration of the study will be approximately up to 21 weeks, including screening period.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be overtly healthy, as determined by medical evaluation.
* Have normal blood pressure, pulse rate, electrocardiogram (ECG), blood and urine laboratory test results that are acceptable for the study.
* Participants must be native Chinese and born in China, where the participant's biological parents and all 4 of the participant's biological grandparents are of Chinese origin.
* Have a body mass index (BMI) within the range of 18.0 to 28.0 kilograms per square meter (kg/m²).
* Have venous access sufficient to allow for blood sampling.

Exclusion Criteria:

* Have known allergies to Lebrikizumab, related compounds, or any components of the formulation.
* Have a significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the investigational medicinal product; or of interfering with the interpretation of data.
* Have a history or presence of psychiatric disorders.
* Have a history or presence of multiple or severe drug allergies.
* Have significant allergies to monoclonal antibodies.
* Show evidence of active or latent TB, human immunodeficiency virus infection ,hepatitis B and C.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 250 mg Lebrikizumab | 500 mg Lebrikizumab | Placebo
Started | 10 | 10 | 4
Received at Least One Dose of Study Drug | 10 | 10 | 4
Completed | 10 | 10 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug.
Groups:
- 250 mg Lebrikizumab: Participants received single dose of 250 mg lebrikizumab administered as SC injection on day 1.
- Total: Total of all reporting groups
Arm/Group | 250 mg Lebrikizumab | 500 mg Lebrikizumab | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 4 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (8.08) | 29.1 (5.95) | 29.0 (6.22) | 30.8 (6.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 7
  Male | 8 | 7 | 2 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 4 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 10 | 10 | 4 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 10 | 10 | 4 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs)
Description: A TEAE is defined as an AE that starts during or after dosing, or starts prior to dosing and increases in severity after dosing. A SAE is defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria listed: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect; is an important medical event that may require medical or surgical intervention to prevent any of the above outcomes.
  A summary of TEAEs, SAEs and other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events section of this record.
Time Frame: Baseline up to 120 days
Population: All enrolled participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | 250 mg Lebrikizumab | 500 mg Lebrikizumab | Placebo
Number analyzed (Participants) | 10 | 10 | 4
participants
  TEAEs | 10 | 10 | 3
  SAEs | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of Lebrikizumab
Description: PK: Cmax of Lebrikizumab is reported.
Time Frame: Day 1: Predose and Days 2, 5, 8, 11, 15, 22, 29, 43, 57, 71, 85, and 120 post dose
Population: All enrolled participants who received at least one dose of lebrikizumab and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per millilitre (µg/mL)
Arm/Group | 250 mg Lebrikizumab | 500 mg Lebrikizumab
Number analyzed (Participants) | 10 | 10
microgram per millilitre (µg/mL) | 26.8 (41.9) | 71.2 (22.1)

3. Secondary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC [0-∞]) of Lebrikizumab
Description: PK: AUC0-∞ of Lebrikizumab is reported.
Time Frame: Day 1: Predose and Days 2, 5, 8, 11, 15, 22, 29, 43, 57, 71, 85, and 120 post dose
Population: All enrolled participants who received at least one dose of lebrikizumab and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*day per milliliter (μg*day/mL)
Arm/Group | 250 mg Lebrikizumab | 500 mg Lebrikizumab
Number analyzed (Participants) | 10 | 10
microgram*day per milliliter (μg*day/mL) | 1130 (42.2) | 2940 (11.2)

4. Secondary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to the Last Measurable Concentration (AUC[0-tlast]) of Lebrikizumab
Description: PK: AUC0-tlast of Lebrikizumab is reported.
Time Frame: Day 1: Predose and Days 2, 5, 8, 11, 15, 22, 29, 43, 57, 71, 85, and 120 post dose
Population: All enrolled participants who received at least one dose of lebrikizumab and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*day/mL
Arm/Group | 250 mg Lebrikizumab | 500 mg Lebrikizumab
Number analyzed (Participants) | 10 | 10
μg*day/mL | 1080 (40.8) | 2800 (11.7)

ADVERSE EVENTS:
Time Frame: Baseline Up to 120 Days
Description: All enrolled participants who received at least one dose of study drug.
Arm/Group | 250 mg Lebrikizumab | 500 mg Lebrikizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/4
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 3/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 250 mg Lebrikizumab (N=10) | 500 mg Lebrikizumab (N=10) | Placebo (N=4)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 3 (4) | 1 (1) | 1 (1)
Noninfective gingivitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Bilirubin conjugated increased (Investigations) | 1 (2) | 3 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (2) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 3 (4) | 1 (1)
Blood triglycerides increased (Investigations) | 2 (5) | 0 (0) | 1 (1)
Blood uric acid increased (Investigations) | 1 (1) | 1 (2) | 0 (0)
Eosinophil count increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 3 (3) | 0 (0)
Urinary occult blood positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Urine ketone body present (Investigations) | 0 (0) | 1 (1) | 0 (0)
Urobilinogen urine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT06243198/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT06243198/SAP_001.pdf